CLINICAL TRIAL: NCT01801527
Title: E-Cuidate: Effectiveness of a Telerehabilitation System in Women Breast Cancer Survivors
Brief Title: Telehealth System to Improve Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Manuel Arroyo Morales, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI10/02749-02764
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Telehealth; Fatigue; Breast cancer; Exercise; Quality of life; Telerehabilitation
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telerehabilitation group (Experimental)
  Interventions: Behavioral: Telerehabilitation group
- Control group (No Intervention): Information about usual care

INTERVENTIONS:
Behavioral: Telerehabilitation group — Interventions will be based on to provide cardiovascular, mobility, strength and stretching exercises through telerehabilitation system
  Arms: Telerehabilitation group

SUMMARY:
Background: Cancer is increasingly viewed as a chronic disease and therefore there is a growing need for long-term treatments. Breast cancer survivors suffer physical impairment after oncology treatment. This impairment reduces quality of life (QoL) and increases the prevalence of conditions associated to unhealthy life-style.

Objective: The overall objective of e-Cuidate telerehabilitation will be to evaluate short and long-term effects telehealth program.

Methods: Seventy-two breast cancer survivors (age range: 18-65 years) will be recruited through oncology and breast units at the Virgen de las Nieves Hospital and San Cecilio Hospital and associations of breast cancer patients in Granada. Patients will be randomized to receive the online rehabilitation group (n=36) or usual care (control) group (n=36). Telerehabilitation group will receive an eight-week online intervention and control group receive recommendations about usual care.

Discussion: The investigators study attempts to increase the level of fitness and reduce musculoskeletal disorders in breast cancer patients through a strategy for care based on telerehabilitation to promote therapeutic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II, or IIIA breast cancer
* Medical clearance of participation
* Without chronic disease or orthopaedic that would interfere with ability to participate in a physical activity program
* Access to Internet
* Basic ability to use the computer or living with a relative who has this ability
* Completion of adjuvant therapy except for hormone therapy
* No history of cancer recurrence
* Have interest in improving lifestyle: fitness/stress level
* Have signed informed consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | Participants will be followed over 8 weeks
  The primary outcome will be assessed with The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0. This questionnaire includes both multi-item scales and single-item measures. These are composed by five functional scales, three symptom scales, a global health status/QoL scale, and six single items. The scores have to be averaged and transformed linearly to obtain a range of score from 0 to 100 where high score meaning a great response level. The European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) which is a breast cancer module of EORTC QLQ-C30 will also be assessed

SECONDARY OUTCOMES:
Algometry | Participants will be followed over 8 weeks
  The pressure pain thresholds (PPTs) will be measured through an electronic algometer (Somedic AB, Farsta, Sweden). PPTs over the C5-C6 zygapophyseal joint, deltoid muscle and tibialis anterior muscle will be assessed bilaterally. The mean of 3 trials will be used for the main analysis
The Visual Analogue Scale (VAS) for pain | Participants will be followed over 8 weeks
  This is a scale for subjective pain estimation that consists of line with a range scored of 0-10 where 0 means 'no pain' and 10 means 'worst pain imaginable'. Participants will have to mark of level of pain that they feel in that moment for both upper limb
Pain | Participants will be followed over 8 weeks
  The Brief Pain Inventory (BPI) short form will be used to assess pain severity and pain interference
Body composition | Participants will be followed over 8 weeks
  Height will be measured. Weight, body mass index, skeletal muscle mass and percentage of body fat will be obtained with bioelectrical impedance analysis (InBody 720; Biospace, Seoul, South Korea)
Physical measurement | Participants will be followed over 8 weeks
  * The Abdominal test (McQuade)
  * Measurement of upper body muscular strength: Handgrip strength will be determined using digital dynamometer (TKK 5101 Grip-D; Takey, Tokyo, Japan)
  * Measurement of back muscle strength: Back muscle strength will be assessed with digital dynamometer (TKK 5002 Back-A; Takey, Tokyo, Japan)
  * Lower body endurance: Multiple sit-to-stand test will be used to assess general lower extremity endurance
Cardiorespiratory fitness | Participants will be followed over 8 weeks
  * The International Fitness Scale (IFIS) will be used to evaluate perceived patients' overall fitness, cardio-respiratory fitness, muscular fitness, speed-agility and flexibility
  * Functional capacity: The 6-minute walk test using a treadmill (H-P-COSMOS for graphics; Germany) will be used to determine the maximum distance (meters) that can be walked in 6 min
Fatigue | Participants will be followed over 8 weeks
  The Piper Fatigue Scale-revised (R-PFS) includes 22 items and four dimensions such as behavioral/severity, affective meaning, sensory and cognitive/mood
Anxiety and depression | Participants will be followed over 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess levels of anxiety and depression. It contains 14 items (7 items for each scale) with 4-point Likert scale
Cognitive function | Participants will be followed over 8 weeks
  * The Trail Making Test (TMT) will be used to assess speed for attention, sequencing, mental flexibility, visual search and motor function. The TMT consists of two parts (A and B)
  * The Auditory Consonant Trigram (ACT) will be used to test short-term memory, divided attention and information-processing capacity in adults
Accelerometry | Participants will be followed over 8 weeks
  Participants will be asked to wear an tri-axial accelerometer (ActiGraph GT3X+, Pensacola, Florida, US) for 8 consecutive days, starting the same day they receive the monitor, and will returned the accelerometers to the researcher 9 days later

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo-Morales, PhD, Principal Investigator — Faculty of Health Sciences. University of Granada
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Spain

REFERENCES:
- [Derived] Galiano-Castillo N, Arroyo-Morales M, Ariza-Garcia A, Fernandez-Lao C, Fernandez-Fernandez AJ, Cantarero-Villanueva I. Factors that Explain the Cancer-Related Insomnia. Breast J. 2017 Jul;23(4):387-394. doi: 10.1111/tbj.12759. Epub 2017 Jan 24. PMID 28117498
- [Derived] Galiano-Castillo N, Ariza-Garcia A, Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Legeren-Alvarez M, Sanchez-Salado C, Del-Moral-Avila R, Arroyo-Morales M. Telehealth system (e-CUIDATE) to improve quality of life in breast cancer survivors: rationale and study protocol for a randomized clinical trial. Trials. 2013 Jun 22;14:187. doi: 10.1186/1745-6215-14-187. PMID 23799886